CLINICAL TRIAL: NCT00465673
Title: A Phase II Study of Liposomal Doxorubicin (Lipo-Dox) in Patients With Brain Metastasis From Breast Cancer
Brief Title: Liposomal Doxorubicin (Lipo-Dox) in Patients With Brain Metastasis From Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: TTY Biopharm (Industry)
Responsible Party: Alex Chang, Johns Hopkins Singapore International Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS 0553
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; brain metastatsis; Lipo-Dox
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Liposomal Doxorubicin — 40mg/m2 over 1 hour infusion for 21 days

SUMMARY:
Primary objective:

To determine the brain response rate of Lipo-Dox in breast cancer patients with brain metastasis

Secondary objectives:

1. To determine the overall objective response rate (ORR)
2. To determine the progression free survival, and duration of objective response
3. To evaluate the overall survival (OS)
4. To assess the safety profiles

DETAILED DESCRIPTION:
This is an open-label, non-comparative phase II clinical trial. Approximately thirty-three patients will be enrolled in order to obtain twenty-nine evaluable subjects who received two cycles of study treatment in Simon's 2-stage optimal design.

Duration of subject involvement: Study treatment should be administered up to disease progression, intolerable toxicity, or consent withdrawal.

Recruitment period: 10 months

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proved breast cancer
* Relapse/recurrent brain metastasis progression after brain radiotherapy
* Presence of brain measurable disease which is defined as at least one brain lesion that can be measured in at least 1 dimension as ³ 20 mm with magnetic resonance image (MRI)
* Prior chemotherapy or hormone therapy for metastatic breast cancer is allowed
* Performance status of ECOG 0, 1, 2
* With normal left ventricular ejection fraction and normal ventricular contractility
* Age 21 years or older
* Life expectancy equal or longer than 3 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior anthracycline-containing chemotherapy with cumulative dose exceed 400mg/m2 doxorubicin or 750 mg/m2 Epirubicin
* Surgery , radiotherapy, hormonal therapy or chemotherapy within 4 weeks prior to entering the study
* Prior liposomal doxorubicin treatment
* Concurrent chemotherapy, radiotherapy, hormonal therapy, or other investigational drug except non-disease related conditions (e.g. insulin for diabetes) during study period
* Other malignancy with exception of curative treated non-melanoma skin cancer or cervical carcinoma in situ within 5 years prior to entering the study
* Brain metastases defined as meninges metastases
* Presence of serious concomitant illness which might be aggravated by study medication:

  * Uncontrolled infection (active serious infections that are not controlled by antibiotics)
  * Active cardiac disease e.g. decompensate myocardial infarction within the 6-month period preceding entry into the study.
  * History of ventricular arrhythmia or congestive heart failure.
* Presence of abnormal left ventricular ejection fraction
* Hematopoietic function as defined below:

  * Hemoglobin<10g/dl
  * ANC< 1,500/uL
  * Platelets<100,000/uL
* Organ function as defined below:

  * Total bilirubin >1.5 × ULN
  * ALT / AST>3 × ULN (>5.0 x ULN if hepatic metastasis)
  * Creatinine >1.5 × ULN
* Mental status is not fit for clinical trial
* Pregnant or breast feeding women, or women of child-bearing potential unless using a reliable and appropriate contraceptive method

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Determine the brain response rate of Lipo-Dox in breast cancer patients with brain metastasis | 3 years

SECONDARY OUTCOMES:
To determine the overall objective response rate | 3 years
To determine the progression free survival, and duration of objective response | 3 years
To evaluate the overall survival | 3 years
To assess the safety profiles | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chang, Principal Investigator — Johns Hopkins SIngapore International Medical Center
Locations (1):
- Johns Hopkins Singapore International Medical Center, Singapore, Singapore